CLINICAL TRIAL: NCT05006599
Title: Study of Nasal Insulin to Fight Forgetfulness (SNIFF) - 3-Week Aptar CPS Device
Brief Title: SNIFF - 3-Week Aptar CPS Device
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: protocol being rewritten and submitted as new study
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00073876
Record Dates: First submitted 2021-07-27; First posted 2021-08-16 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-03

CONDITIONS: Mild Cognitive Impairment; Cognitive Impairment; Alzheimer Disease, Early Onset
Keywords: Intranasal Delivery of Insulin; Cognitive Testing; Nasal Insulin
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither participants or site personnel will know which drug intervention (insulin or placebo) is being administered. Exceptions will be the Study Nurse who is directly involved in preparing the insulin or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Humulin® R U-100 (Experimental): Twenty randomly assigned participants with Alzheimer's disease or mild cognitive impairment will receive intranasal administrations of Humulin® R U-100 (40 IU) four times daily for 3 weeks.
  Interventions: Drug: Insulin (Humulin® R U-100); Device: Aptar Pharma CPS Intranasal Delivery Device
- Placebo (Placebo Comparator): Twenty randomly assigned participants with Alzheimer's disease or mild cognitive impairment will receive intranasal administrations of placebo (insulin diluent) four times daily for 3 weeks.
  Interventions: Drug: Placebo; Device: Aptar Pharma CPS Intranasal Delivery Device

INTERVENTIONS:
Drug: Insulin (Humulin® R U-100) — Participants will administer 40 IU of Humulin® U-100 insulin four times per day with an intranasal delivery device.
  Arms: Humulin® R U-100
Drug: Placebo — Participants will administer placebo (insulin diluent) four times per day with an intranasal delivery device.
  Other Names: Insulin Diluent
  Arms: Placebo
Device: Aptar Pharma CPS Intranasal Delivery Device — Participants will be assigned to receive Humulin® insulin or placebo administered through the Aptar Pharma CPS intranasal delivery device.

SUMMARY:
The SNIFF 3-Week Aptar Device study will involve using a device to administer insulin or placebo through each participant's nose or intra-nasally. Insulin is a hormone that is produced in the body. It works by lowering levels of glucose (sugar) in the blood. This study is measuring how much insulin the device delivers. In addition, this study will look at the effects of insulin or placebo administered intra-nasally using an intranasal delivery device on memory, blood, and cerebrospinal fluid (CSF).

DETAILED DESCRIPTION:
The proposed study will examine whether an intranasal delivery device can be used by adults with preclinical Alzheimer's disease (cognitively normal but with abnormal brain levels of the hallmark peptide Aβ) to reliably deliver insulin or placebo four times daily over a 4 week period. We will also examine effects of treatment on cognition, CSF biomarkers, and cerebral perfusion. If successful, information gained from the study will inform the design of future Phase III trials of intranasal insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 to 85 (inclusive)
2. Fluent in English
3. Cognitively normal or diagnosis of amnestic mild cognitive impairment (aMCI) or mild Alzheimer's disease (AD)
4. Amyloid positive by positron emission tomography (PET) or cerebrospinal fluid (CSF) criteria
5. Stable medical condition for 3 months prior to screening visit
6. Stable medications for 4 weeks prior to the screening and study visits (exceptions may be made on a case by case basis by the study physician)
7. Clinical laboratory values must be within normal limits or, if abnormal, must be judged to be clinically insignificant by the study physician

Exclusion Criteria:

1. A diagnosis of dementia other than Alzheimer's disease (AD)
2. History of a clinically significant stroke
3. Current evidence or history in past two years of epilepsy, head injury with loss of consciousness, any major psychiatric disorder including psychosis, major depression, bipolar disorder
4. Diabetes (type I or type II) insulin-dependent and non-insulin-dependent diabetes mellitus
5. Current or past regular use of insulin or any other anti-diabetic medication within 2 months of screening visit
6. History of seizure within past five years
7. Pregnancy or possible pregnancy
8. Use of anticoagulants
9. Residence in a skilled nursing facility at screening
10. Use of an investigational agent within two months of screening visit
11. Regular use of alcohol, narcotics, anticonvulsants, anti-parkinsonian medications, or any other exclusionary medications (exceptions may be made on a case by case basis by the study physician)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Prescribed Dose Taken | Week 4
  Participant self-reported medication adherence information will be calculated by study staff on a 0%-100% scale. A score below 80% indicates low medication adherence and a score of 80% or higher indicates high medication adherence.

SECONDARY OUTCOMES:
Change in the Preclinical Alzheimer Cognitive Composite 5 (PACC5) Z-Score | Baseline to Week 8
  Cognition will be measured using the PACC5 scale, which includes the free/cued selective reminding test, delayed paragraph recall, digit-symbol substitution, mini mental state score, and the category fluency task. The PACC5 is a composite score comprised of measures of global cognition, memory, and executive function. The score reflects an averaged z-score, with higher scores indicating better cognitive performance.
Change in the 14-item Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog 14) Score | Baseline to Week 8
  A psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis. A higher score indicates more impairment. Scores from the original portion of the test range from 0 (best) to 65 (worse), and are added to the mean of the words not immediately recalled (max of 10) and the number of items not recalled after a delay (ranging from 0-10) all total the maximum score of 85. A positive change indicates cognitive worsening.
Change in Cerebrospinal Fluid (CSF) Insulin Levels | Baseline to Week 8
  Measurement of the levels of insulin in cerebrospinal fluid (CSF) after being delivered with the intranasal delivery device. This will help to determine the ability of the intranasal delivery device to increase levels of insulin in CSF.
Change in amyloid β-peptide (Aβ) 40 (Aβ40) in Cerebrospinal Fluid (CSF) | Baseline to Week 8
  Cerebrospinal fluid (CSF) samples will be used to measure the levels of amyloid β-peptide (Aβ) 40. CSF Aβ40 is a key Alzheimer's disease (AD) biomarker that reflects pathological aggregation of amyloid in the brain.
Change in amyloid β-peptide (Aβ) 42 (Aβ42) in Cerebrospinal Fluid (CSF) | Baseline to Week 8
  Cerebrospinal fluid (CSF) samples will be used to measure the levels of amyloid β-peptide (Aβ) 42. CSF Aβ42 is a key Alzheimer's disease (AD) biomarker that reflects pathological aggregation of amyloid in the brain.
Change in Cerebrospinal Fluid (CSF) Levels of Total Tau | Baseline to Week 8
  Cerebrospinal fluid (CSF) samples will be used to measure the levels of total tau protein in the brain to assess impact on brain tau as a relevant Alzheimer's Disease (AD) biomarker.
Change in Cerebrospinal Fluid (CSF) Levels of Phospho-Tau 181 | Baseline to Week 8
  Cerebrospinal fluid (CSF) samples will be used to measure the levels of phospho-tau 181 protein in the brain to assess impact on brain tau as a relevant Alzheimer's Disease (AD) biomarker.
Change in Cerebrospinal Fluid (CSF) Levels of Phospho-Tau 217 | Baseline to Week 8
  Cerebrospinal fluid (CSF) samples will be used to measure the levels of phospho-tau 217 protein in the brain to assess impact on brain tau as a relevant Alzheimer's Disease (AD) biomarker.

OTHER OUTCOMES:
Change in Quick Dementia Rating Scale (QDRS) Score | Baseline to Week 8
  The QDRS (Galvin, 2015) is a clinical scale that rates the severity of dementia as absent, questionable, mild, moderate, or severe (Clinical Dementia Rating score of 0, 0.5, 1, 2, or 3, respectively). The score assesses six domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. At Screening the QDRS global score will be used for eligibility purposes. For all other administrations, the 6 domain scores will be summed to get the QDRS Sum of Boxes (SB) score. Sum of boxes score ranges from 0-100 with a high score meaning more severe dementia.
Change in Patient Health Questionnaire (PHQ-9) Score | Baseline to Week 8
  The Patient Health Questionnaire (PHQ-9) is a 9-item, validated measure of depression severity. Respondents indicate how bothered by problems they are on a scale from 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 27, where higher scores indicate more severe depression.
Change in Generalized Anxiety Disorder scale-7 (GAD-7) Score | Baseline to Week 8
  Changes in anxiety will be measured using the Generalized Anxiety Disorder Scale (GAD-7), which contains 7 items with total scores ranging from 0 to 21. Scores of 5, 10, and 15 are cut-offs for mild, moderate, and severe anxiety, respectively.
Change in PROMIS Sleep Disturbance Questionnaire Score | Baseline to Week 8
  A questionnaire to assess self-reported quality of general sleep and sleep disturbance. Each item on the form is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Change in the Alzheimer's Disease Cooperative Study Activities of Daily Living Scale for Mild Cognitive Impairment (ADCS-ADL-MCI) | Baseline to Week 8
  An interview-based assessment of information provided by the study partner (informant). The total scores based on 18 items on the scale range from 0 to 53 with lower scores representing greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Baker H, Spencer RF. Transneuronal transport of peroxidase-conjugated wheat germ agglutinin (WGA-HRP) from the olfactory epithelium to the brain of the adult rat. Exp Brain Res. 1986;63(3):461-73. doi: 10.1007/BF00237470. PMID 3758265
- [Background] Baker LD, Cross DJ, Minoshima S, Belongia D, Watson GS, Craft S. Insulin resistance and Alzheimer-like reductions in regional cerebral glucose metabolism for cognitively normal adults with prediabetes or early type 2 diabetes. Arch Neurol. 2011 Jan;68(1):51-7. doi: 10.1001/archneurol.2010.225. Epub 2010 Sep 13. PMID 20837822
- [Background] Balin BJ, Broadwell RD, Salcman M, el-Kalliny M. Avenues for entry of peripherally administered protein to the central nervous system in mouse, rat, and squirrel monkey. J Comp Neurol. 1986 Sep 8;251(2):260-80. doi: 10.1002/cne.902510209. PMID 3782501
- [Background] Benedict C, Hallschmid M, Hatke A, Schultes B, Fehm HL, Born J, Kern W. Intranasal insulin improves memory in humans. Psychoneuroendocrinology. 2004 Nov;29(10):1326-34. doi: 10.1016/j.psyneuen.2004.04.003. PMID 15288712
- [Background] Benedict C, Kern W, Schultes B, Born J, Hallschmid M. Differential sensitivity of men and women to anorexigenic and memory-improving effects of intranasal insulin. J Clin Endocrinol Metab. 2008 Apr;93(4):1339-44. doi: 10.1210/jc.2007-2606. Epub 2008 Jan 29. PMID 18230654
- [Background] Born J, Lange T, Kern W, McGregor GP, Bickel U, Fehm HL. Sniffing neuropeptides: a transnasal approach to the human brain. Nat Neurosci. 2002 Jun;5(6):514-6. doi: 10.1038/nn849. No abstract available. PMID 11992114
- [Background] Broadwell RD, Balin BJ. Endocytic and exocytic pathways of the neuronal secretory process and trans-synaptic transfer of wheat germ agglutinin-horseradish peroxidase in vivo. J Comp Neurol. 1985 Dec 22;242(4):632-50. doi: 10.1002/cne.902420410. PMID 2418083
- [Background] Cavanna AE, Trimble MR. The precuneus: a review of its functional anatomy and behavioural correlates. Brain. 2006 Mar;129(Pt 3):564-83. doi: 10.1093/brain/awl004. Epub 2006 Jan 6. PMID 16399806
- [Background] Chiu SL, Chen CM, Cline HT. Insulin receptor signaling regulates synapse number, dendritic plasticity, and circuit function in vivo. Neuron. 2008 Jun 12;58(5):708-19. doi: 10.1016/j.neuron.2008.04.014. PMID 18549783
- [Background] Craft S, Baker LD, Montine TJ, Minoshima S, Watson GS, Claxton A, Arbuckle M, Callaghan M, Tsai E, Plymate SR, Green PS, Leverenz J, Cross D, Gerton B. Intranasal insulin therapy for Alzheimer disease and amnestic mild cognitive impairment: a pilot clinical trial. Arch Neurol. 2012 Jan;69(1):29-38. doi: 10.1001/archneurol.2011.233. Epub 2011 Sep 12. PMID 21911655
- [Background] Craft S, Peskind E, Schwartz MW, Schellenberg GD, Raskind M, Porte D Jr. Cerebrospinal fluid and plasma insulin levels in Alzheimer's disease: relationship to severity of dementia and apolipoprotein E genotype. Neurology. 1998 Jan;50(1):164-8. doi: 10.1212/wnl.50.1.164. PMID 9443474
- [Background] Craft S, Watson GS. Insulin and neurodegenerative disease: shared and specific mechanisms. Lancet Neurol. 2004 Mar;3(3):169-78. doi: 10.1016/S1474-4422(04)00681-7. PMID 14980532
- [Background] De Felice FG, Vieira MN, Bomfim TR, Decker H, Velasco PT, Lambert MP, Viola KL, Zhao WQ, Ferreira ST, Klein WL. Protection of synapses against Alzheimer's-linked toxins: insulin signaling prevents the pathogenic binding of Abeta oligomers. Proc Natl Acad Sci U S A. 2009 Feb 10;106(6):1971-6. doi: 10.1073/pnas.0809158106. Epub 2009 Feb 2. PMID 19188609
- [Background] Fishel MA, Watson GS, Montine TJ, Wang Q, Green PS, Kulstad JJ, Cook DG, Peskind ER, Baker LD, Goldgaber D, Nie W, Asthana S, Plymate SR, Schwartz MW, Craft S. Hyperinsulinemia provokes synchronous increases in central inflammation and beta-amyloid in normal adults. Arch Neurol. 2005 Oct;62(10):1539-44. doi: 10.1001/archneur.62.10.noc50112. PMID 16216936
- [Background] Francis GJ, Martinez JA, Liu WQ, Xu K, Ayer A, Fine J, Tuor UI, Glazner G, Hanson LR, Frey WH 2nd, Toth C. Intranasal insulin prevents cognitive decline, cerebral atrophy and white matter changes in murine type I diabetic encephalopathy. Brain. 2008 Dec;131(Pt 12):3311-34. doi: 10.1093/brain/awn288. Epub 2008 Nov 16. PMID 19015157 (Retraction: PMID 24860127 Brain. 2014 Jun;137(Pt 6):e283)
- [Background] Frolich L, Blum-Degen D, Bernstein HG, Engelsberger S, Humrich J, Laufer S, Muschner D, Thalheimer A, Turk A, Hoyer S, Zochling R, Boissl KW, Jellinger K, Riederer P. Brain insulin and insulin receptors in aging and sporadic Alzheimer's disease. J Neural Transm (Vienna). 1998;105(4-5):423-38. doi: 10.1007/s007020050068. PMID 9720972
- [Background] Galasko D, Bennett D, Sano M, Ernesto C, Thomas R, Grundman M, Ferris S. An inventory to assess activities of daily living for clinical trials in Alzheimer's disease. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S33-9. PMID 9236950
- [Background] Gasparini L, Gouras GK, Wang R, Gross RS, Beal MF, Greengard P, Xu H. Stimulation of beta-amyloid precursor protein trafficking by insulin reduces intraneuronal beta-amyloid and requires mitogen-activated protein kinase signaling. J Neurosci. 2001 Apr 15;21(8):2561-70. doi: 10.1523/JNEUROSCI.21-08-02561.2001. PMID 11306609
- [Background] Gil-Bea FJ, Solas M, Solomon A, Mugueta C, Winblad B, Kivipelto M, Ramirez MJ, Cedazo-Minguez A. Insulin levels are decreased in the cerebrospinal fluid of women with prodomal Alzheimer's disease. J Alzheimers Dis. 2010;22(2):405-13. doi: 10.3233/JAD-2010-100795. PMID 20847404
- [Background] Hallschmid M, Benedict C, Schultes B, Born J, Kern W. Obese men respond to cognitive but not to catabolic brain insulin signaling. Int J Obes (Lond). 2008 Feb;32(2):275-82. doi: 10.1038/sj.ijo.0803722. Epub 2007 Sep 11. PMID 17848936
- [Background] Hong M, Lee VM. Insulin and insulin-like growth factor-1 regulate tau phosphorylation in cultured human neurons. J Biol Chem. 1997 Aug 1;272(31):19547-53. doi: 10.1074/jbc.272.31.19547. PMID 9235959
- [Background] Hughes CP, Berg L, Danziger WL, Coben LA, Martin RL. A new clinical scale for the staging of dementia. Br J Psychiatry. 1982 Jun;140:566-72. doi: 10.1192/bjp.140.6.566. PMID 7104545
- [Background] Illum L. Nasal drug delivery: new developments and strategies. Drug Discov Today. 2002 Dec 1;7(23):1184-9. doi: 10.1016/s1359-6446(02)02529-1. PMID 12547019
- [Background] Kern W, Born J, Schreiber H, Fehm HL. Central nervous system effects of intranasally administered insulin during euglycemia in men. Diabetes. 1999 Mar;48(3):557-63. doi: 10.2337/diabetes.48.3.557. PMID 10078556
- [Background] Kristensson K, Olsson Y. Uptake of exogenous proteins in mouse olfactory cells. Acta Neuropathol. 1971;19(2):145-54. doi: 10.1007/BF00688493. No abstract available. PMID 5126829
- [Background] Kupila A, Sipila J, Keskinen P, Simell T, Knip M, Pulkki K, Simell O. Intranasally administered insulin intended for prevention of type 1 diabetes--a safety study in healthy adults. Diabetes Metab Res Rev. 2003 Sep-Oct;19(5):415-20. doi: 10.1002/dmrr.397. PMID 12951650
- [Background] Lee CC, Kuo YM, Huang CC, Hsu KS. Insulin rescues amyloid beta-induced impairment of hippocampal long-term potentiation. Neurobiol Aging. 2009 Mar;30(3):377-87. doi: 10.1016/j.neurobiolaging.2007.06.014. Epub 2007 Aug 10. PMID 17692997
- [Background] Minoshima S, Frey KA, Foster NL, Kuhl DE. Preserved pontine glucose metabolism in Alzheimer disease: a reference region for functional brain image (PET) analysis. J Comput Assist Tomogr. 1995 Jul-Aug;19(4):541-7. doi: 10.1097/00004728-199507000-00006. PMID 7622680
- [Background] Minoshima S, Koeppe RA, Frey KA, Kuhl DE. Anatomic standardization: linear scaling and nonlinear warping of functional brain images. J Nucl Med. 1994 Sep;35(9):1528-37. PMID 8071705
- [Background] Morris JC, Ernesto C, Schafer K, Coats M, Leon S, Sano M, Thal LJ, Woodbury P. Clinical dementia rating training and reliability in multicenter studies: the Alzheimer's Disease Cooperative Study experience. Neurology. 1997 Jun;48(6):1508-10. doi: 10.1212/wnl.48.6.1508. PMID 9191756
- [Background] Petersen RC, Doody R, Kurz A, Mohs RC, Morris JC, Rabins PV, Ritchie K, Rossor M, Thal L, Winblad B. Current concepts in mild cognitive impairment. Arch Neurol. 2001 Dec;58(12):1985-92. doi: 10.1001/archneur.58.12.1985. PMID 11735772
- [Background] Pontiroli AE, Alberetto M, Secchi A, Dossi G, Bosi I, Pozza G. Insulin given intranasally induces hypoglycaemia in normal and diabetic subjects. Br Med J (Clin Res Ed). 1982 Jan 30;284(6312):303-6. doi: 10.1136/bmj.284.6312.303. PMID 6800439
- [Background] Reger MA, Watson GS, Frey WH 2nd, Baker LD, Cholerton B, Keeling ML, Belongia DA, Fishel MA, Plymate SR, Schellenberg GD, Cherrier MM, Craft S. Effects of intranasal insulin on cognition in memory-impaired older adults: modulation by APOE genotype. Neurobiol Aging. 2006 Mar;27(3):451-8. doi: 10.1016/j.neurobiolaging.2005.03.016. Epub 2005 Jun 16. PMID 15964100
- [Background] Reger MA, Watson GS, Green PS, Baker LD, Cholerton B, Fishel MA, Plymate SR, Cherrier MM, Schellenberg GD, Frey WH 2nd, Craft S. Intranasal insulin administration dose-dependently modulates verbal memory and plasma amyloid-beta in memory-impaired older adults. J Alzheimers Dis. 2008 Apr;13(3):323-31. doi: 10.3233/jad-2008-13309. PMID 18430999
- [Background] Reger MA, Watson GS, Green PS, Wilkinson CW, Baker LD, Cholerton B, Fishel MA, Plymate SR, Breitner JC, DeGroodt W, Mehta P, Craft S. Intranasal insulin improves cognition and modulates beta-amyloid in early AD. Neurology. 2008 Feb 5;70(6):440-8. doi: 10.1212/01.WNL.0000265401.62434.36. Epub 2007 Oct 17. PMID 17942819
- [Background] Rivera EJ, Goldin A, Fulmer N, Tavares R, Wands JR, de la Monte SM. Insulin and insulin-like growth factor expression and function deteriorate with progression of Alzheimer's disease: link to brain reductions in acetylcholine. J Alzheimers Dis. 2005 Dec;8(3):247-68. doi: 10.3233/jad-2005-8304. PMID 16340083
- [Background] Sakane T, Akizuki M, Taki Y, Yamashita S, Sezaki H, Nadai T. Direct drug transport from the rat nasal cavity to the cerebrospinal fluid: the relation to the molecular weight of drugs. J Pharm Pharmacol. 1995 May;47(5):379-81. doi: 10.1111/j.2042-7158.1995.tb05814.x. PMID 7494186
- [Background] Sano M, Raman R, Emond J, Thomas RG, Petersen R, Schneider LS, Aisen PS. Adding delayed recall to the Alzheimer Disease Assessment Scale is useful in studies of mild cognitive impairment but not Alzheimer disease. Alzheimer Dis Assoc Disord. 2011 Apr-Jun;25(2):122-7. doi: 10.1097/WAD.0b013e3181f883b7. PMID 20921876
- [Background] Selkoe DJ. Soluble oligomers of the amyloid beta-protein impair synaptic plasticity and behavior. Behav Brain Res. 2008 Sep 1;192(1):106-13. doi: 10.1016/j.bbr.2008.02.016. Epub 2008 Feb 17. PMID 18359102
- [Background] Shipley MT. Transport of molecules from nose to brain: transneuronal anterograde and retrograde labeling in the rat olfactory system by wheat germ agglutinin-horseradish peroxidase applied to the nasal epithelium. Brain Res Bull. 1985 Aug;15(2):129-42. doi: 10.1016/0361-9230(85)90129-7. PMID 3840049
- [Background] Stockhorst U, de Fries D, Steingrueber HJ, Scherbaum WA. Insulin and the CNS: effects on food intake, memory, and endocrine parameters and the role of intranasal insulin administration in humans. Physiol Behav. 2004 Oct 30;83(1):47-54. doi: 10.1016/j.physbeh.2004.07.022. PMID 15501490
- [Background] Thorne RG, Emory CR, Ala TA, Frey WH 2nd. Quantitative analysis of the olfactory pathway for drug delivery to the brain. Brain Res. 1995 Sep 18;692(1-2):278-82. doi: 10.1016/0006-8993(95)00637-6. PMID 8548316
- [Background] Thorne RG, Pronk GJ, Padmanabhan V, Frey WH 2nd. Delivery of insulin-like growth factor-I to the rat brain and spinal cord along olfactory and trigeminal pathways following intranasal administration. Neuroscience. 2004;127(2):481-96. doi: 10.1016/j.neuroscience.2004.05.029. PMID 15262337
- [Background] Townsend M, Mehta T, Selkoe DJ. Soluble Abeta inhibits specific signal transduction cascades common to the insulin receptor pathway. J Biol Chem. 2007 Nov 16;282(46):33305-33312. doi: 10.1074/jbc.M610390200. Epub 2007 Sep 13. PMID 17855343
- [Background] Weiss P, Holland Y. Neuronal dynamics and axonal flow, ii. The olfactory nerve as model test object. Proc Natl Acad Sci U S A. 1967 Feb;57(2):258-64. doi: 10.1073/pnas.57.2.258. No abstract available. PMID 16591462
- [Background] Worsley KJ, Evans AC, Marrett S, Neelin P. A three-dimensional statistical analysis for CBF activation studies in human brain. J Cereb Blood Flow Metab. 1992 Nov;12(6):900-18. doi: 10.1038/jcbfm.1992.127. PMID 1400644
- [Background] Zhao L, Teter B, Morihara T, Lim GP, Ambegaokar SS, Ubeda OJ, Frautschy SA, Cole GM. Insulin-degrading enzyme as a downstream target of insulin receptor signaling cascade: implications for Alzheimer's disease intervention. J Neurosci. 2004 Dec 8;24(49):11120-6. doi: 10.1523/JNEUROSCI.2860-04.2004. PMID 15590928
- [Background] Zhao WQ, Townsend M. Insulin resistance and amyloidogenesis as common molecular foundation for type 2 diabetes and Alzheimer's disease. Biochim Biophys Acta. 2009 May;1792(5):482-96. doi: 10.1016/j.bbadis.2008.10.014. Epub 2008 Nov 5. PMID 19026743
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171